CLINICAL TRIAL: NCT05343780
Title: A Phase II, Randomized, Double Blind, Placebo-Controlled Clinical Trial to Investigate the Anti-oxidant Activity of Heptex in Patients With Apparent Risk Factors of Nonalcoholic Steatohepatitis (NASH)
Brief Title: Clinical Trial to Investigate the Anti-oxidant Activity of Heptex in Patients With Apparent Risk Factors of NASH
Acronym: PHYLLANTEX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Natural Wellness Egypt (Industry)
Collaborators: Ain Shams University (Other); National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NW_PHYLLANTEX_17052018
Record Dates: First submitted 2019-05-15; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo (Rice bran) in 2 capsules size 1, administered PO TID on empty stomach with plenty of water.
  Interventions: Other: Rice bran
- Heptex-low dose (Experimental): Low dose The contents of one capsule of Heptex is equally distributed and inserted into 2 capsules size 1, administered PO TID on empty stomach with plenty of water.
  Interventions: Drug: Heptex
- Heptex-high dose (Experimental): High dose The contents of two capsule of Heptex is equally distributed and inserted into 2 capsules size 1, administered PO TID on empty stomach with plenty of water.
  Interventions: Drug: Heptex

INTERVENTIONS:
Drug: Heptex — Dukung Anak 200 mg + Milk thistle 100 mg
  Arms: Heptex-high dose; Heptex-low dose
Other: Rice bran — Placebo
  Arms: Placebo

SUMMARY:
A Phase II, Randomized, Double Blind, Placebo-Controlled Clinical Trial to Investigate the Anti-oxidant Activity of Heptex in Patients with Apparent Risk Factors of Nonalcoholic Steatohepatitis (NASH)

DETAILED DESCRIPTION:
This is a phase II, randomized, double blind placebo-controlled, three-arm, parallel-group, intervention clinical trial evaluating anti-oxidant activity of Heptex; a herbal medicinal product of Aerial Parts of Phyllanthus niruri (Dukung Anak) and Fruits of Silybum marianum (Milk Thistle) in patients with apparent risk factors of NASH.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged between 18 and 65 years.
2. Both male and female patients who have childbearing potential must agree to practice an acceptable method of birth control during the study and for at least 6 months after the cessation of treatment; such contraceptive methods must include at least one barrier method.
3. Controlled Attenuation Parameter (CAP)-confirmed hepatic steatosis.
4. Patients with elevated serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels but less than 2.5 times the upper limit of the normal range.
5. Liver fibrosis stage F1-F2 as diagnosed by the FibroScan liver stiffness measurement of 5-10 kPa.
6. Liver condition according the following criteria;

   * Serum albumin > 3 g/dl
   * INR < 2
   * No ascites on ultrasound
   * No documented or suspected hepatic encephalopathy
7. Willing to stop any other liver support and hepatoprotective medications throughout study duration.
8. Able and willing to provide written informed consent.
9. Able and willing to complete all study visits and procedures, including compliance with the requirements and restrictions listed in the consentform.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with BMI > 40 Kg/m2 or BMI < 18.5 Kg/m2.
3. Serum creatinine > 1.5 x ULN OR creatinine clearance (GFR) < 60 mL/minute.
4. Platelet count < 75,000/mm3.
5. Uncontrolled diabetes mellitus as evident by HbA1c ≥ 8.5%.
6. Patients who are currently receiving Thiazolidinediones.
7. Patients with ischemic heart disease (IHD).
8. History of parenteral nutrition.
9. History of liver transplant.
10. Viral hepatitis, drug-induced liver injury, metabolic liver disease or auto-immune liver disease.
11. Liver cancer or serum alpha-fetoprotein (AFP) >100ng/ml. Patients with an AFP between 50 and 100ng/ml may be included as long as a liver ultrasound within 3 months of screening, or at screening, shows no evidence of potential hepatocellular cancer.
12. Use of drugs known to induce steatosis (valproate, amiodarone or prednisone) or to affect body weight and carbohydrate metabolism.
13. Use of drugs known to alter liver enzymes.
14. Allergy or allergic history to any of the drug components.
15. History of alcohol abuse as assessed by the investigator within the past 2 years, or an alcohol use pattern that may interfere with the patient's study compliance. Patients must have abstained from alcohol for at least 6 months prior to study start.
16. Patients with history of clinically-significant illness or any other major medical disorder that may interfere with subject treatment, assessment, or compliance with the protocol.
17. Receipt of an investigational drug within 6 months prior to screening, or active enrolment in another investigational medication or device trial.
18. Patients with any chronic illness or prior treatment which in the opinion of the investigator should preclude participation in the trial.
19. Inability to understand and cooperate with the investigators or to give valid consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
explore the anti-oxidant activity of Heptex | 36 weeks
  assessed by the change in serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels in patients with apparent risk factors of NASH.

SECONDARY OUTCOMES:
explore the hepatoprotective effect of Heptex | 36 weeks
  assessed by the change in Fibrosis score (F0 to F1: 2 to 7 kPa, F2: 7.5 to 10 kPa, F3: 10 to 14 kPa, F4: 14 kPa or higher) and by the occurrence of hepatic complications.

OTHER OUTCOMES:
To explore the lipid-lowering effect of Heptex | 36 weeks
  To explore the lipid-lowering effect of Heptex as assessed by the change in lipid profile.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - National Hepatology & Tropical Medicine Research Instistute, Cairo
  - Tropical Medicine Department, Faculty of Medicine, Ain Shams University, Cairo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shaker MK, Hassany M, Eysa B, Adel A, Zidan A, Mohamed S. The activity of a herbal medicinal product of Phyllanthus niruri and Silybum marianum powdered extracts (Heptex(R)) in patients with apparent risk factors for nonalcoholic steatohepatitis: a phase II, multicentered, randomized, double-blind, placebo-controlled clinical trial. BMC Complement Med Ther. 2025 Jan 9;25(1):8. doi: 10.1186/s12906-024-04692-y. PMID 39789561

DOCUMENTS (1):
  • Study Protocol (2019-12-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT05343780/Prot_000.pdf